CLINICAL TRIAL: NCT00319657
Title: Total Lymphoid Irradiation, Anti-Thymocyte Globulin and Purified Donor CD34+ and T-Cell Transfusion in HLA-Matched Living Donor Kidney Transplantation
Brief Title: Kidney and Blood Stem Cell Transplantation That Eliminates Requirement for Immunosuppressive Drugs
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Samuel Strober, Chair of Study, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 367; P01HL075462-02 (NIH)
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Immune Tolerance
Keywords: Kidney Transplantation; Blood Stem Cell Transplantation
MeSH Terms: interventions — Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: Combined hematopoietic stem cell and kidney transplantation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immune tolerance, kidney transplantation (Experimental): Intervention: Participants will receive hematopoietic cell transplantation and Total lymphoid irradiation. The intervention is intended to induce immune tolerance in HLA-matched living donor kidney transplantation, to allow withdrawal of the immunosuppressive drugs. Immune tolerance is achieved through the development of donor/recipient mixed chimerism following combined kidney and hematopoietic stem cell transplantation from the living donor.
  Interventions: Biological: Hematopoietic cell transplantation; Radiation: Total lymphoid irradiation

INTERVENTIONS:
Biological: Hematopoietic cell transplantation — Transplantation of hematopoietic stem cells from the living donor.
Radiation: Total lymphoid irradiation — Total lymphoid irradiation is used as part of the conditioning regimen for the hematopoietic stem cell transplant.

SUMMARY:
The Stanford Medical Center Program in Multi-Organ Transplantation and the Division of Bone Marrow Transplantation are enrolling patients into a research study to determine if blood stem cells injected after kidney transplantation, in combination with lymphoid irradiation ,will change the immune system such that immunosuppressive drugs can be completely withdrawn. Patients must have a healthy, completely human leukocyte antigen (HLA)-matched brother or sister as the organ and stem cell donor.

One to two months before kidney transplant surgery, blood stem cells will be removed from the donor and the cells will be frozen. After transplant surgery, the recipient will receive radiation and anti-T cell antibody treatments for two weeks to prepare for injection of the stem cells. The stem cells will be injected at the end of the two-week treatment. If the stem cells persist in the recipient, immunosuppressive drugs will be gradually reduced until they are withdrawn completely at least six months after transplantation. Patients will be followed in the Stanford clinics for transplant patients. Patients who live outside of the San Francisco Bay Area must remain near Stanford for six weeks after transplant surgery.

DETAILED DESCRIPTION:
The purpose of this study is to determine the proportion of patients that can be withdrawn completely from immunosuppressive drugs while maintaining normal function of HLA-matched living related donor kidney transplants. Fifteen participants will be conditioned with total lymphoid irradiation (TLI) and rabbit anti-thymocyte globulin (ATG), and given an infusion of donor "mobilized" blood mononuclear cells prior to transplantation.

This is a single-center, open-label study in adult renal transplant patients. Fifteen patients will receive TLI, ATG, and an infusion of CD34+ selected G-CSF mobilized blood cells combined with a fixed number (1x10^6) of CD3+ T cells from the same mobilized blood cell source. Patients will receive a one-month course of mycophenolate mofetil and a six to 12 month tapering course of cyclosporine that will be discontinued at six months. At serial timepoints (1) graft function will be monitored, (2) chimerism will be measured in recipient white blood cell subsets, (3) mixed lymphocyte response (MLR) assays of peripheral blood mononuclear cells against donor and third party cells will be performed, and (4) protocol biopsies of the graft will be obtained. An attempt will be made to discontinue cyclosporine at six months if (1) chimerism is detectable for at least 180 days after CD34+ and CD3+ cell infusion, (2) there is stable graft function without clinical rejection episodes, and (3) there is lack of histologic rejection on protocol biopsies. In the proposed study, patients will be given a target dose of 8-10x10^6 CD34+ cells/kg and 1x10^6 CD3+ cells/kg because sustained chimerism may be necessary for sustained tolerance to the graft.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant performed at Stanford University Medical Center
* Have an HLA-matched sibling donor
* No known contraindication to administration of rabbit ATG or radiation
* Willing to use a reliable form of contraception for at least 24 months following transplantation

Exclusion Criteria:

* Previous treatment with rabbit ATG or a known allergy to rabbit proteins
* History of cancer, other than non-melanoma skin cancer
* Pregnant or breastfeeding
* HIV, Hepatitis B, or Hepatitis C infection
* Previous organ transplant
* Leukopenia (white blood cell count less than 3000/mm³)
* Thrombocytopenia (platelet count less than 100,000/mm³)
* cPRA>80%

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2004-07; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Discontinuation of maintenance immunosuppressive drugs | Measured at 12 months
  Study subjects are discontinued from immunosuppressive drugs as they have achieved immune tolerance at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Strober, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual Patient Data will not be shared

REFERENCES:
- [Background] Strober S, Benike C, Krishnaswamy S, Engleman EG, Grumet FC. Clinical transplantation tolerance twelve years after prospective withdrawal of immunosuppressive drugs: studies of chimerism and anti-donor reactivity. Transplantation. 2000 Apr 27;69(8):1549-54. doi: 10.1097/00007890-200004270-00005. PMID 10836360
- [Background] Millan MT, Shizuru JA, Hoffmann P, Dejbakhsh-Jones S, Scandling JD, Grumet FC, Tan JC, Salvatierra O, Hoppe RT, Strober S. Mixed chimerism and immunosuppressive drug withdrawal after HLA-mismatched kidney and hematopoietic progenitor transplantation. Transplantation. 2002 May 15;73(9):1386-91. doi: 10.1097/00007890-200205150-00005. PMID 12023614
- [Result] Scandling JD, Busque S, Shizuru JA, Engleman EG, Strober S. Induced immune tolerance for kidney transplantation. N Engl J Med. 2011 Oct 6;365(14):1359-60. doi: 10.1056/NEJMc1107841. No abstract available. PMID 21991976
- [Result] Scandling JD, Busque S, Dejbakhsh-Jones S, Benike C, Sarwal M, Millan MT, Shizuru JA, Lowsky R, Engleman EG, Strober S. Tolerance and withdrawal of immunosuppressive drugs in patients given kidney and hematopoietic cell transplants. Am J Transplant. 2012 May;12(5):1133-45. doi: 10.1111/j.1600-6143.2012.03992.x. Epub 2012 Mar 8. PMID 22405058
- [Derived] Jensen KP, Hongo DA, Ji X, Zheng P, Pawar R, Wu TH, Busque S, Scandling JD, Shizuru JA, Lowsky R, Shori A, Dutt S, Waters J, Saraswathula A, Baker J, Tamaresis JS, Lavori P, Negrin R, Maecker H, Engleman EG, Meyer E, Strober S. Development of immunosuppressive myeloid cells to induce tolerance in solid organ and hematopoietic cell transplant recipients. Blood Adv. 2021 Sep 14;5(17):3290-3302. doi: 10.1182/bloodadvances.2020003669. PMID 34432869